CLINICAL TRIAL: NCT05201001
Title: An Early Phase Randomized Trial of APX005M in BRCAwt Patients With Recurrent Ovarian Cancer
Brief Title: APX005M in Patients With Recurrent Ovarian Cancer
Acronym: APX005M
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IMP provider company (Apexigen) is sold, thus both IMP and grant is terminated
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: Belgian Gynaecological Oncology Group (Other); GSO Global Clinical Research BV (Other); The Central and Eastern European Gynecologic Oncology Group (Other); Swiss GO Trial Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-OV64/NSGO-CTU-SOLERO
Record Dates: First submitted 2021-07-09; First posted 2022-01-21 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — sotigalimab; Radiotherapy; Carboplatin; 1-dodecylpyridoxal

STUDY DESIGN:
Intervention Model Description: randomised, open-label, three arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): Carboplatin AUC = 5, IV day 1 and pegylated liposomal doxorubicin (PLD) 30 mg/m , IV day1 q4 wks
  Total:6 cycles or until progressive disease or unacceptable toxicity.
  Interventions: Drug: APX005M
- APX005M (Experimental): Carboplatin AUC = 5, IV day 1 combined with pegylated liposomal doxorubicin (PLD) 30 mg/m , IV day1 q4 wks APX005M 0.3 mg/kg, days 1 & 15 IV q4 wks x concomitant with chemotherapy
  Total:6 cycles or until progressive disease or unacceptable toxicity.
  Interventions: Drug: APX005M
- APX005M+RT (Experimental): Carboplatin AUC = 5, IV day 1 combined with pegylated liposomal doxorubicin (PLD) 30 mg/m , IV day1 q4 wks APX005M 0.3 mg/kg, days 1 & 15 IV q4 wks x concomitant with chemotherapy External beam radiation therapy; a dose of 0.5 Gy per fraction, administered as single fractions prior to APX005M administration; days 1 & 15 q4 wks x 6 cycles. Maximum 24 wks of therapy; total dose 6 Gy.
  Total:6 cycles or until progressive disease or unacceptable toxicity.
  Interventions: Drug: APX005M

INTERVENTIONS:
Drug: APX005M — adding immunotherapy with or without radiation therapy to chemotherapy. Low dose radiation therapy is to sensitise tumour cells to immunotherapy.
  Other Names: Radiation therapy; carboplatin and PLD

SUMMARY:
The overall objective is to demonstrate preliminary efficacy of APX005M-carboplatin-PLD and APX005M-radiotherapy-carboplatin-PLD combinations as treatment for relapsed BRCAwt ovarian cancer patients, where platinum combination therapy is an option.

DETAILED DESCRIPTION:
The rationale for integrating immunotherapy with chemotherapy is based on preclinical studies, which have shown, that chemotherapy induces immunogenic cell death leading to increased recognition of the tumor by the immune system. Carboplatin is shown to inhibit PD-L2 expression, thereby limiting immunosuppression by both dendritic cells and tumor cells. Paclitaxel decreases the percentage of CD4+ and FoxP3+ regulatory T cells (Tregs) and reduces their cytokine production without disrupting the function of its effector counterpart (CD4+ and FoxP3 effector T (Teff) cells). Several trials have shown effect of checkpoint inhibition following chemotherapy and radiotherapy, most notably in the PACIFIC trial in stage III NSCLC [63]. We therefore hypothesize, that the proposed combined therapies will yield improved clinical effect in this patient population.

The hypotheses in this study is, that the CD-40 agonist APX005M with or without radiotherapy, and in combination with platinum-doublet chemotherapy, will provide the necessary immune activation and serve as a basis for increased clinical effect of the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form prior to any study-specific evaluation.
2. Histologically diagnosed epithelial ovarian, fallopian tube or primary peritoneal cancer.
3. Radiological or histological confirmation of relapse disease ≥ 6 month after last chemotherapy
4. Known BRCAwt
5. Have completed at least one line of platinum-containing chemotherapy (maximum three previous lines of therapy are permitted). Earlier PARPi treatment permitted
6. Must have measurable or evaluable disease according to RESIST 1.1.
7. Baseline biopsy: Tissue biopsy for submission to central laboratory prior to study treatment should be from a newly obtained metastatic biopsy, if there is a lesion suitable for biopsy. If a metastatic biopsy is not feasible, or patient is unwilling to provide new biopsy, archival tissue samples should be submitted. Archival tissue sample from metastatic site is preferred; however, archival tissue sample of primary tumor is acceptable.
8. Must consent to undergo mandatory tumor biopsy of at least one metastatic site at baseline and at day 84 ( 7). Biopsy at day 84 ( 7) is only applicable if surgery is not performed. -

Exclusion Criteria:

1. Previous immunotherapy (for example anti-PD-1/L1).
2. Other malignancy unless curatively treated with no evidence of disease for ≥ 3years, except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) and stage 1 grade 1 endometrial carcinoma.
3. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or subjects with congenital long QT syndrome.
4. Subjects with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML. Page 48 af 128 ENGOT-OV64/NSGO-CTU-SOLERO EudraCT: 2020-005990-29 Final Version 1.0, 06. July 2021
5. Subjects with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Subjects with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
6. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Subjects who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) or physiologic replacement doses (i.e. prednisone 5 - 7.5 mg/day) for adrenal insufficiency may be enrolled in the study. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
7. Prior radiation therapy.
8. Planned concomitant therapy with any other anticancer therapy
9. Conditions requiring ongoing therapy with antibiotics
10. History of any arterial thromboembolic event within 3 months prior to first dose of APX005M
11. Active coagulopathy
12. Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation
13. History of organ transplant
14. Major surgery or significant traumatic injury within 4 weeks prior to first dose of study drugs
15. Pregnant or breastfeeding women.
16. Subjects with a known hypersensitivity to any of the excipients of the product.
17. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy, except alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    1. Subjects with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Lead Principal Investigator (PI) of the respective collaborative group
    2. Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with study drugs may be included only after consultation with the Lead PI of the respective collaborative group.
18. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Subjects with vitiligo or alopecia
    2. Subjects with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement Page 49 af 128 ENGOT-OV64/NSGO-CTU-SOLERO EudraCT: 2020-005990-29 Final Version 1.0, 06. July 2021
    3. Any chronic skin condition that does not require systemic therapy
    4. Subjects without active disease in the last 5 years may be included, but only after consultation with the Lead PI of the respective collaborative group.
    5. Subjects with celiac disease controlled by diet alone
19. Subjects considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, recent (within 3 months), uncontrolled major seizure disorder, serious chronic gastrointestinal conditions associated with diarrhea, interstitial lung disease or any psychiatric disorder/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the Subject to give written informed consent.
20. Immunocompromised subjects, e.g. subjects who are known to be serologically positive for human immunodeficiency virus (HIV).
21. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg)), hepatitis C.

    Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
22. Receipt of live attenuated vaccine within 30 days prior to the first dose of Investigational Product (IP). Note: Subjects, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP. COVID-19 vaccination must be performed minimum 7 days prior to first dose of APX005M. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 0 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate according to RECIST at 12 weeks of treatment | 18 months
  To evaluate the preliminary efficacy of APX005M-carboplatin-PLD and APX005M radiotherapycarboplatin-PLD combinations

SECONDARY OUTCOMES:
Adverse events | 18 months
  To evaluate adverse events, safety & feasibility of the two combinations

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, Study Chair — NSGO-CTU
Locations (1):
- NSGO-CTU, Copenhagen, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
NSGO-CTU can be contacted